CLINICAL TRIAL: NCT02816697
Title: Implementation of a System-level Tobacco Treatment Intervention in Thoracic Oncology
Brief Title: Implementation of a System-level Tobacco Treatment Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mary E. Cooley, Phd, Mary E. Cooley MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-208
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Lung Cancer
Keywords: Smoking Habits
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cease-Aim 1 (Active Comparator): * Cease Implementation
  * 100 Patients after CEASE Implementation
    * Exit Interview and Tobacco Use Survey
  Interventions: Other: CEASE
- Pre Cease Implementation Aim 2 (Active Comparator): 50 Current or former smokers (3 months +/-2 month) patients in usual care (before CEASE implementation)
  * Tobacco Use Survey (Baseline,1- 6 Months)
  * Biochemical verification
  Interventions: Other: Usual Care Tobacco Treatment Services
- After Cease Implementation Aim 2 (Experimental): 50 Current or former smokers (3 months +/-2 month)
  * Tobacco Use Survey (Baseline,1- 6 Months)
  * Biochemical verification
  Interventions: Other: CEASE
- Usual Care-Aim 1 (Active Comparator): Usual Care Tobacco Treatment Services
  * 100 patients in usual care
  * Exit Interview and Tobacco Use Survey
  Interventions: Other: Usual Care Tobacco Treatment Services
- Clinician and Staff Survey (No Intervention): - Interview clinicians and support staff (40)

INTERVENTIONS:
Other: CEASE — * Clinical and Community Effort Against Secondhand Smoke Exposure (CEASE)
  * CEASE is a system-level intervention that integrates tobacco-use screening, cessation assistance, and referral to outside services into routine visits
  Arms: After Cease Implementation Aim 2; Cease-Aim 1
Other: Usual Care Tobacco Treatment Services
  Arms: Pre Cease Implementation Aim 2; Usual Care-Aim 1

SUMMARY:
The proposed study plans to adapt and study the implementation and effectiveness of integrating Clinical and Community Effort Against Secondhand smoke Exposure (CEASE) into the thoracic oncology setting using mixed methods.

DETAILED DESCRIPTION:
In particular the study aims to see if participants are asked about their smoking status and what services are offered if someone indicates being a former or current smoker. Findings from this study will help improve a standard of care at this clinic and allow us to understand what type of tobacco treatment services are preferred by patients.

* Adaption of CEASE will entail exit interviews with patients and individual interviews with clinical staff to identify and address facilitators and barriers to the implementation process.
* Effectiveness of CEASE will be measured through questionnaires & biochemical verification of smoking status using a pre-test/post-test study design before (usual care)and after implementation (CEASE)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Have an actual or potential diagnosis of thoracic malignancy
* Able to read and write in English.
* Current or recent former smoker (defined as having smoked within past 6 months)
* Must have an active telephone number.

Exclusion Criteria:

* Former smoker greater than 6 months.
* Have any of the below conditions needing immediate medical intervention

  * Hypercalcemia causing lethargy and confusion,
  * Acute respiratory distress
  * Dehydration
  * Hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation Rate | 6 Months
  Biochemical verification of smoking cessation

SECONDARY OUTCOMES:
Documentation of tobacco treatment | 2 months after CEASE
  Assess documentation of smoking assessment and provision of treatment ( medication and referral for behavioral counseling)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Cooley, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No